CLINICAL TRIAL: NCT02105961
Title: Study MEA117113: Mepolizumab vs. Placebo as Add-on Treatment for Frequently Exacerbating COPD Patients Characterized by Eosinophil Level
Brief Title: Efficacy and Safety of Mepolizumab as an Add-on Treatment in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 117113
Record Dates: First submitted 2014-04-03; First posted 2014-04-07 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; exacerbations; SB240563; mepolizumab; eosinophils
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Each subject will receive 100 mg mepolizumab SC injection every 4 weeks (13 administrations during 52 week treatment period) along with their baseline standard of care COPD medication
  Interventions: Drug: Mepolizumab
- Arm 2 (Experimental): Each subject will receive 300 mg mepolizumab SC injection every 4 weeks (13 administrations during 52 week treatment period) along with their baseline standard of care COPD medication
  Interventions: Drug: Mepolizumab
- Arm 3 (Experimental): Each subject will receive placebo (0.9percent sodium chloride) SC injection every 4 weeks (13 administrations during 52 week treatment period) their baseline standard of care COPD medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mepolizumab — Humanised IgG antibody (IgG1, kappa) with human heavy and light chain frameworks, provided as a lyophilised cake in sterile vial. Vial to be reconstituted with Sterile Water for Injection, just prior to use.
  Arms: Arm 1; Arm 2
Drug: Placebo — Sterile 0.9percent sodium chloride solution
  Arms: Arm 3

SUMMARY:
This is a multi-centered, randomized, placebo-controlled, double-blind, parallel group, trial evaluating 2 doses of mepolizumab against placebo given every 4 weeks through subcutaneous (SC) injection. In severe COPD subjects, sputum eosinophils levels are elevated to similar levels as those seen in severe asthmatics. It is hypothesized that the reduction of eosinophils with mepolizumab in COPD subjects would translate into a reduction of COPD exacerbations. The study will evaluate the efficacy and safety of mepolizumab, in subjects who are at or above the baseline blood eosinophil count of at least 150 cells/microliters who exacerbate despite regular use of maximal tolerated therapy, appropriate for severe COPD subjects, in the 12 months prior to study start. In total, 660 subjects will be randomized in 1:1:1 ratio to receive mepolizumab 300 mg, mepolizumab 100mg, or placebo administered SC. The total duration of subject participation will be approximately 62 weeks, consisting of a 1 to 2 week screening period, 52-week treatment period and 8-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis: Subjects with a clinically documented history of COPD for at least 1 year in accordance with the following definition by the American Thoracic Society/European Respiratory Society
* Severity of COPD: Subjects must present with the following: a measured pre and post-salbutamol Forced expiratory volume in one second/ Forced vital capacity (FEV1/FVC) ratio of <0.70 at Visit 1 to confirm the diagnosis of COPD; a measured post-salbutamol FEV1> 20 percent and <=80 percent of predicted normal values calculated using National Health and Nutrition Examination Survey (NHANES) III reference equations at Visit 1
* History of exacerbations: A well documented history (e.g., medical record verification) in the 12 months prior to Visit 1 of ; at least two moderate COPD exacerbations. Moderate is defined as the use of systemic corticosteroids (intramuscular (IM), intravenous, or oral) and/or treatment with antibiotics or; at least one severe COPD exacerbation. Severe is defined as having required hospitalization. Note: At least one exacerbation must have occurred while the subject was taking Inhaled corticosteroid (ICS) plus long acting beta2-agonist (LABA) plus long acting muscarinic antagonist (LAMA). Prior use of antibiotics alone does not qualify as a moderate exacerbation unless the use was specifically for the treatment of worsening symptoms of COPD.
* Concomitant COPD therapy: A well documented requirement for optimized standard of care background therapy that includes Inhaled corticosteroid (ICS) plus 2 additional COPD medications (i.e., triple therapy) for the 12 months prior to Visit 1 and meets the following criteria: Immediately prior to Visit 1, minimum of 3 months of use of an; Inhaled corticosteroid at a dose >= 500 micrograms (mcg)/day fluticasone propionate dose equivalent plus; LABA and LAMA.

For subjects who are not continually maintained on ICS plus LABA plus LAMA for the entire 12 months prior to Visit 1 use of following is allowed (but not in the 3 months immediately prior to Visit 1); inhaled corticosteroid at a dose >=500 mcg/day fluticasone propionate dose equivalent plus; a LABA or a LAMA and; use of at least one other class of COPD medication (i.e., phosphodiesterase-4-inhibitors, methylxanthines, or a combination of short acting beta2-agonist and short acting muscarinic antagonist).

* Informed Consent: Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Gender: Male or Eligible Female; To be eligible for entry into the study females of child bearing potential must commit to consistent and correct use of an acceptable method of birth control from the time of consent, for the duration of the trial, and for 4 months after last study drug administration.
* Age: At least 40 years of age at Visit 1
* Smoking status: Subject with confirmed COPD are eligible to participate independent of their smoking status and smoking history, i.e. current smokers, never smokers or ex-smokers can be enrolled into the study. Current smokers are defined as those with a history of cigarette smoking of >=10 pack-years [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Former smokers are defined as those who meet the definition of a current smoker but have stopped smoking for at least 6 months prior to Visit 1. Never smokers are those that do not meet the definition of a current or former smoker.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Subjects with Asthma: Current and Former Smokers: Subjects with a current diagnosis of asthma (those with a prior history are eligible if they meet inclusion criteria for a current diagnosis of COPD); Never-Smokers: Subjects with any history of asthma.
* Other respiratory disorders: The investigator must judge that COPD is the primary diagnosis accounting for the clinical manifestations of the lung disease. Subjects with alpha1-antitrypsin deficiency as the underlying cause of COPD are excluded. Also, excluded are subjects with active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, primary pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases. Subjects are also excluded if maintenance use of bi-level positive airway pressure is required for the treatment of respiratory disorder.
* COPD stability: Subjects with pneumonia, exacerbation, lower respiratory infection within the 4 weeks prior to Visit 1.
* Lung resection: Subjects with lung volume reduction surgery within the 12 months prior to Visit 1.
* Pulmonary rehabilitation program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Oxygen: Subjects receiving treatment with oxygen more than 4.0 liters/minute (L/min). While breathing supplemental oxygen, subjects should demonstrate an oxyhemoglobin saturation greater than or equal to 89 percent.
* 12-lead Electrocardiography (ECG) finding: An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1, if considered to be clinically significant by the Investigator. 12-lead ECGs will be over-read by a centralized independent cardiologist to assist in consistent evaluation of subject eligibility. Results from the 12-lead ECG over-read must be received prior to assessing eligibility at Visit 2.
* Unstable or life threatening cardiac disease: Subjects with any of the following would be excluded: Myocardial infarction or unstable angina in the last 6 months ; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months ; New York Heart Association (NYHA) Class IV Heart failure
* Other diseases/abnormalities: Subjects with (historical or) current evidence of clinically significant, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Eosinophilic disease: Subjects with other conditions that could lead to elevated eosinophils such as Hypereosinophilic syndromes including Eosinophilic Granulomatosis with Polyangiitis (EGPA, also known as Churg-Strauss Syndrome), or Eosinophilic Esophagitis.
* Parasitic infection: Subjects with a pre-existing helminthes infestation within 6 months prior to Visit 1 are also excluded.
* Malignancy: A current malignancy or previous history of cancer in remission for less than 12 months prior to Visit 1 (Subjects that had localized carcinoma of the skin or cervix which was resected for cure will not be excluded). South Korea subjects with a diagnosis of malignancy within 5 years of Visit 1 are excluded.
* Immunodeficiency: A known immunodeficiency (e.g. human immunodeficiency virus HIV), other than that explained by the use of corticosteroids taken for COPD.
* Liver disease: Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, and known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Chronic stable hepatitis B and C are acceptable if subject otherwise meets entry criteria (e.g., presence of hepatitis B surface antigen or positive hepatitis C test result within 3 months of screening)
* Monoclonal antibodies: Subjects who have received any monoclonal antibody within 5 half-lives of Visit 1.
* Investigational medications: Subjects who have received an investigational drug within 30 days of Visit 1, or within 5 drug half-lives of the investigational drug, whichever is longer (this also includes investigational formulations of a marketed product).
* Hypersensitivity: Subjects with a known allergy or intolerance to another monoclonal antibody or biologic including history of anaphylaxis to another biologic
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete study related materials.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Drug or alcohol abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Previous participation: Subjects who have previously participated in any study of mepolizumab.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.

Randomization Criteria

In order to be randomized to study drug the subject must meet the following randomization criteria at Visit 2:

* Blood eosinophils: Documented elevated peripheral blood eosinophil count of >=300 cells/microliter within the past 12 months prior to Visit 1; OR A peripheral baseline blood eosinophil count of >=150 cells/microliter from haematology conducted at Visit 1
* Electronic Diary Compliance: Compliance with completion of the eDiary defined as completion of all questions on 5 or more days out of the 7 days immediately preceding Visit 2.
* 12-lead ECG: No evidence of an abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1 as indicated on the over-read provided by the centralized independent cardiologist. Subjects with a QT interval corrected with Fridericia's formulas (QTcF)>=450 msec are not eligible. For subjects with a QRS interval >=120msec, those with QTcF>=480 msec are not eligible. Specific ECG findings that preclude subject eligibility are listed in the protocol.
* Abnormal chest X-ray (or Computerized Tomography [CT] scan): No chest X-ray (or CT scan) that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. If a chest X-ray or CT scan is not available within 6 months prior to Visit 1, then a chest X-ray must be taken at Visit 1 and the results reviewed prior to randomization. For sites in Germany: If a chest X-ray (or CT scan) within 6 months prior to Screening (Visit 1) is not available, the subject will not be eligible for the study.
* Laboratory abnormality: No evidence of clinically significant abnormality in the haematological, biochemical, or urinalysis screen at Visit 1, as judged by the investigator.
* Hepatitis B: Subjects who are HBsAg positive or HBcAb positive must not have a HBV DNA level >=2000 International Units (IU)/millilitre (mL).
* Liver function test: Subjects must meet the following based on results from sample taken at Visit 1: Alanine aminotransferase (ALT) <2x ULN (upper limit of normal); Alkaline Phosphatase (Alk Phos) <=2x ULN; Bilirubin <=1.5x ULN (isolated bilirubin>1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent)
* Pregnancy: No subjects who are pregnant or breastfeeding. Subjects should not be enrolled if they plan to become pregnant during the time of study participation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (139):
- United States (34):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Broomfield, Colorado
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Adairsville, Georgia
  - GSK Investigational Site, Duluth, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Bowling Green, Kentucky
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Oaks, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Morgantown, West Virginia
- Argentina (7):
  - GSK Investigational Site, Bahía Blanca, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Berazategui
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (3):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Murdoch, Western Australia
- Canada (6):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Chile (4):
  - GSK Investigational Site, Talca, Maule Region
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Denmark (4):
  - GSK Investigational Site, Aarhus C
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, København NV
  - GSK Investigational Site, Odense C
- Germany (12):
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Japan (20):
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Shimane
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Netherlands (10):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Horn
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Sittard-geleen
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Zutphen
- Romania (9):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Codlea
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Focşani
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Timișoara
- Slovakia (5):
  - GSK Investigational Site, Humenné
  - GSK Investigational Site, Poprad
  - GSK Investigational Site, Spišská Nová Ves
  - GSK Investigational Site, Šaľa
  - GSK Investigational Site, Vráble
- South Korea (9):
  - GSK Investigational Site, Anyang-Si Gyeonggi-do
  - GSK Investigational Site, Bucheon City, Gyenggi-do
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Wonju-si, Kanwon-do
- Taiwan (4):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan County
- Ukraine (6):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolayiv
  - GSK Investigational Site, Vinnytsia
- United Kingdom (6):
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Pavord ID, Chapman KR, Bafadhel M, Sciurba FC, Bradford ES, Schweiker Harris S, Mayer B, Rubin DB, Yancey SW, Paggiaro P. Mepolizumab for Eosinophil-Associated COPD: Analysis of METREX and METREO. Int J Chron Obstruct Pulmon Dis. 2021 Jun 16;16:1755-1770. doi: 10.2147/COPD.S294333. eCollection 2021. PMID 34163157
- [Derived] Condreay LD, Gao C, Bradford E, Yancey SW, Ghosh S. No genetic associations with mepolizumab efficacy in COPD with peripheral blood eosinophilia. Respir Med. 2019 Aug;155:26-28. doi: 10.1016/j.rmed.2019.07.004. Epub 2019 Jul 5. PMID 31295674
- [Derived] Roger JH, Bratton DJ, Mayer B, Abellan JJ, Keene ON. Treatment policy estimands for recurrent event data using data collected after cessation of randomised treatment. Pharm Stat. 2019 Jan;18(1):85-95. doi: 10.1002/pst.1910. Epub 2018 Nov 8. PMID 30406948
- [Derived] Pavord ID, Chanez P, Criner GJ, Kerstjens HAM, Korn S, Lugogo N, Martinot JB, Sagara H, Albers FC, Bradford ES, Harris SS, Mayer B, Rubin DB, Yancey SW, Sciurba FC. Mepolizumab for Eosinophilic Chronic Obstructive Pulmonary Disease. N Engl J Med. 2017 Oct 26;377(17):1613-1629. doi: 10.1056/NEJMoa1708208. Epub 2017 Sep 11. PMID 28893134
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic obstructive pulmonary disease (COPD) with frequent exacerbations, on high dose inhaled corticosteroid (ICS)-based triple inhaled maintenance therapy were included. Participants were randomized to receive mepolizumab (100 or 300 milligrams [mg]) or placebo by subcutaneous (SC) injection every 4 weeks for up to 52 weeks.
Pre-assignment Details: A total of 674 participants were randomized and received at least one dose of study treatment and were included in the modified intent to treat (mITT) population. One participant randomized to the mepolizumab 300 mg group was withdrawn without receiving study treatment.
Groups:
- Placebo: Eligible participants were randomized to and received placebo by SC injection every 4 weeks for up to 52 weeks in addition to their standard of care (SoC) therapy. Salbutamol metered dose inhaler (MDI) was issued for use as rescue medication throughout the study.
- Mepolizumab 100 mg SC: Eligible participants were randomized to and received mepolizumab 100 mg by SC injection every 4 weeks for up to 52 weeks in addition to their SoC therapy. Salbutamol MDI was issued for use as rescue medication throughout the study.
- Mepolizumab 300 mg SC: Eligible participants were randomized to and received mepolizumab 300 mg by SC injection every 4 weeks for up to 52 weeks in addition to their SoC therapy. Salbutamol MDI was issued for use as rescue medication throughout the study.
Period: Overall Study
Arm/Group | Placebo | Mepolizumab 100 mg SC | Mepolizumab 300 mg SC
Started | 226 | 223 | 225
Completed Investigational Product (IP) | 170 | 196 | 183
Not Completed IP | 56 | 27 | 42
Withdrew IP Due to: Adverse Event | 27 | 9 | 25
Withdrew IP Due to: Stopping Criteria | 1 | 1 | 0
Withdrew IP Due to: Lack of Efficacy | 6 | 2 | 2
Withdrew IP Due to: Protocol Deviation | 2 | 0 | 1
Withdrew IP Due to: Lost to Follow-up | 1 | 1 | 1
Withdrew IP Due to: Physician Decision | 2 | 3 | 1
Withdrew IP Due to: Withdrawal by Subj. | 16 | 11 | 11
Withdrew IP Due to: Site Closed | 1 | 0 | 1
Completed | 185 | 206 | 195
Not Completed | 41 | 17 | 30
Not completed — Adverse Event | 18 | 7 | 13
Not completed — Lack of Efficacy | 3 | 0 | 3
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Physician Decision | 3 | 3 | 2
Not completed — Withdrawal by Subject | 15 | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eligible participants were randomized to and received placebo by SC injection every 4 weeks for up to 52 weeks in addition to their SoC therapy. Salbutamol MDI was issued for use as rescue medication throughout the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Mepolizumab 100 mg SC | Mepolizumab 300 mg SC | Total
Number analyzed (Participants) | 226 | 223 | 225 | 674
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (8.64) | 64.8 (9.06) | 64.8 (8.96) | 65.1 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 91 | 67 | 228
  Male | 156 | 132 | 158 | 446
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: Asian-Central/South Asian Heritage | 0 | 0 | 1 | 1
  Race customized: Asian-East Asian Heritage | 25 | 26 | 26 | 77
  Race customized: Asian-Japanese Heritage | 14 | 13 | 13 | 40
  Race customized: Asian-South East Asian Heritage | 3 | 2 | 1 | 6
  Race customized: Black or African American | 2 | 4 | 2 | 8
  Race customized: White-White/Caucasian/European Heritage | 182 | 178 | 182 | 542

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate or Severe Exacerbations
Description: Moderate exacerbations are defined as clinically significant exacerbations that require treatment with oral/systemic corticosteroids and/or antibiotics. Severe exacerbations are defined as clinically significant exacerbations that require in-patient hospitalization (>=24 hours) or result in death. Moderate and severe exacerbations occurring from the start of investigational product (IP) up to the Week 52 visit, including exacerbations reported after early discontinuation from IP by participants who remained in the study, were included in the analysis. The analysis was performed on the modified intent-to-treat (mITT) Population (all randomized participants who received at least one dose of study treatment).
Time Frame: From randomization to Week 52
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Moderate/severe exacerbations per year
Groups:
- Mepolizumab 300 mg SC: Eligible participants were randomized to and received mepolizumab 100 mg by SC injection every 4 weeks for up to 52 weeks in addition to their SoC therapy. Salbutamol MDI was issued for use as rescue medication throughout the study.
Arm/Group | Placebo | Mepolizumab 100 mg SC | Mepolizumab 300 mg SC
Number analyzed (Participants) | 226 | 223 | 225
Moderate/severe exacerbations per year | 1.49 [1.29 to 1.72] | 1.19 [1.02 to 1.38] | 1.27 [1.09 to 1.48]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.068, Negative binomial model — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Rate ratio (Mepolizumab 100/Placebo) = 0.80, 95% CI 2-sided [0.65 to 0.98] — Analysis using a negative binomial model with covariates of treatment, geographic region, no. of moderate/severe exacerbations in previous year, Baseline percent predicted FEV1, smoking status and offset of log (time in on- and off- treatment period)
Statistical Analysis 2: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.034, Negative binomial model — Unadjusted p-value; Rate ratio (Mepolizumab 100/Placebo) = 0.80, 95% CI 2-sided [0.65 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.140, Negative binomial model — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Rate ratio (Mepolizumab 300/Placebo) = 0.86, 95% CI 2-sided [0.70 to 1.05] — Analysis using a negative binomial model with covariates of treatment, geographic region, no. of moderate/severe exacerbations in previous year, Baseline percent predicted FEV1, smoking status and offset of log (time in on- and off- treatment period
Statistical Analysis 4: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.140, Negative binomial model — Unadjusted p-value; Rate ratio (Mepolizumab 300/Placebo) = 0.86, 95% CI 2-sided [0.70 to 1.05] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Time to First Moderate/Severe Exacerbation
Description: Kaplan Meier estimates of the probability of a moderate or severe exacerbation are expressed as the percentage of participants with an exacerbation over time (by Week 8, 16, 24, 32, 40, 48, 52). Analysis of time to first moderate/severe exacerbation was performed on the mITT population and included exacerbations reported on-treatment and those reported after early discontinuation from IP by participants who remained in the study.
Time Frame: From randomization to Week 52
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Mepolizumab 100 mg SC | Mepolizumab 300 mg SC
Number analyzed (Participants) | 226 | 223 | 225
Percentage of participants
  Week 8 | 22.6 [17.7 to 28.6] | 22.9 [17.9 to 29.0] | 18.3 [13.8 to 24.0]
  Week 16 | 40.7 [34.6 to 47.5] | 36.0 [30.0 to 42.6] | 29.0 [23.5 to 35.4]
  Week 24 | 51.1 [44.6 to 57.8] | 42.4 [36.2 to 49.2] | 36.7 [30.8 to 43.4]
  Week 32 | 58.3 [51.8 to 64.9] | 46.1 [39.8 to 52.9] | 44.9 [38.7 to 51.7]
  Week 40 | 62.3 [55.8 to 68.7] | 50.8 [44.4 to 57.6] | 51.8 [45.4 to 58.6]
  Week 48 | 64.2 [57.8 to 70.6] | 55.5 [49.1 to 62.2] | 58.3 [51.9 to 64.9]
  Week 52 | 66.7 [60.2 to 73.1] | 57.9 [51.5 to 64.5] | 58.8 [52.4 to 65.3]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.140, Cox Proportional Hazards Model — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Hazard Ratio(Mepolizumab 100/Placebo) = 0.82, 95% CI 2-sided [0.64 to 1.04] — Analysis performed using a Cox Proportional Hazards Model with covariates of treatment, geographic region, number of moderate/severe exacerbations in previous year, Baseline percent predicted FEV1 and smoking status
Statistical Analysis 2: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.103, Cox Proportional Hazards Model — Unadjusted p-value; Hazard Ratio (Mepolizumab/Placebo) = 0.82, 95% CI 2-sided [0.64 to 1.04] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.140, Cox Proportional Hazards Model — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Hazard Ratio (Mepolizumab 300/Placebo) = 0.77, 95% CI 2-sided [0.60 to 0.97] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.030, Cox Proportional Hazards Model — Unadjusted p-value; Hazard Ratio (Mepolizumab 300/Placebo) = 0.77, 95% CI 2-sided [0.60 to 0.97] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Rate of COPD Exacerbations Requiring Emergency Department (ED) Visits and/or Hospitalizations (Hosp)
Description: COPD exacerbations requiring an ED visit and/or hosp occurring from the start of IP up to the Week 52 visit, including exacerbations reported after early discontinuation from IP by participants who remained in the study, were included in the analysis. This analysis was performed on the mITT population.
Time Frame: From randomization to Week 52
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations requiring ED/hosp per year
Arm/Group | Placebo | Mepolizumab 100 mg SC | Mepolizumab 300 mg SC
Number analyzed (Participants) | 226 | 223 | 225
Exacerbations requiring ED/hosp per year | 0.28 [0.20 to 0.40] | 0.17 [0.11 to 0.25] | 0.23 [0.16 to 0.33]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.140, Negative binomial model — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Rate ratio (Mepolizumab 100/Placebo) = 0.59, 95% CI 2-sided [0.35 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.042, Negative binomial model — Unadjusted p-value; Rate ratio (Mepolizumab 100/Placebo) = 0.59, 95% CI 2-sided [0.35 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.447, Negative binomial model — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Rate ratio (Mepolizumab 300/Placebo) = 0.83, 95% CI 2-sided [0.51 to 1.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.447, Negative binomial model — Unadjusted p-value; Rate ratio (Mepolizumab 300/Placebo) = 0.83, 95% CI 2-sided [0.51 to 1.34] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Mean Total St. George's Respiratory Questionnaire (SGRQ) Score
Description: The SGRQ for COPD is a 40-item questionnaire derived from the original SGRQ , designed to measure health impairment by addressing the frequency of respiratory symptoms and current state of the participant. SGRQ Total Scores range from 0 to 100 with higher scores indicating worse health-related quality of life and reductions indicating improvement. The Baseline value will be the last measurement collected prior to the first dose of investigational product.Change from Baseline is calculated as the post-dose visit value minus the Baseline value. Mean change from Baseline in SGRQ score at Week 52 has been presented.
Time Frame: Baseline and Week 52
Population: mITT Population. Participants analyzed represents those with a Baseline and at least one post-Baseline assessment, and with no missing covariates.
Measure: Least Squares Mean (Standard Error); unit: Score on SGRQ scale
Arm/Group | Placebo | Mepolizumab 100 mg SC | Mepolizumab 300 mg SC
Number analyzed (Participants) | 218 | 218 | 219
Score on SGRQ scale | -3.1 (0.98) | -5.0 (0.95) | -3.3 (0.96)
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.447, Mixed Model Repeated Measures Analysis — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Mean difference(Mepolizumab 100-Placebo) = -1.8, 95% CI 2-sided [-4.5 to 0.8] — Analysis performed using mixed model repeated measures with covariates of Baseline SGRQ total score, geographic region, smoking status, treatment and visit, plus interaction terms for visit by Baseline and visit by treatment group
Statistical Analysis 2: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.180, Mixed Model Repeated Measures Analysis — Unadjusted p-value; Mean difference(Mepolizumab 100-Placebo) = -1.8, 95% CI 2-sided [-4.5 to 0.8] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.926, Mixed Model Repeated Measures Analysis — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Mean difference(Mepolizumab 300-Placebo) = -0.1, 95% CI 2-sided [-2.8 to 2.6] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.926, Mixed Model Repeated Measures Analysis — Unadjusted p-value; Mean difference(Mepolizumab 300-Placebo) = -0.1, 95% CI 2-sided [-2.8 to 2.6] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Mean COPD Assessment Test (CAT) Score
Description: The CAT is an 8-item questionnaire developed for use in routine clinical practice to measure the health status of participants with COPD. Each question is assessed on a 6-point scale ranging from 0 (no impairment) to 5 (maximum impairment) with the CAT score ranging from 0-40. Higher scores indicate greater disease impact with reductions indicating improvement. The Baseline value will be the last measurement collected prior to the first dose of investigational product. Change from Baseline is calculated as the post-dose visit value minus the Baseline value. Mean change from Baseline in CAT score at Week 52 has been presented.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Score on CAT scale
Arm/Group | Placebo | Mepolizumab 100 mg SC | Mepolizumab 300 mg SC
Number analyzed (Participants) | 222 | 216 | 219
Score on CAT scale | -0.4 (0.42) | -1.6 (0.42) | -0.8 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.926, Mixed Model Repeated Measures Analysis — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Mean difference(Mepolizumab 100-Placebo) = -1.1, 95% CI 2-sided [-2.3 to 0.0] — Analysis performed using mixed model repeated measures with covariates of Baseline CAT score, geographic region, smoking status, treatment and visit, plus interaction terms for visit by Baseline and visit by treatment group
Statistical Analysis 2: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.055, Mixed Model Repeated Measures Analysis — Unadjusted p-value; Mean difference(Mepolizumab 100-Placebo) = -1.1, 95% CI 2-sided [-2.3 to 0.0] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.926, Mixed Model Repeated Measures Analysis — Adjusted p-value; Family wise type I error controlled within each endpoint using a Hochberg testing procedure; Mean difference(Mepolizumab 300-Placebo) = -0.4, 95% CI 2-sided [-1.5 to 0.8] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mepolizumab 300 mg SC; Test type: Superiority; p = 0.547, Mixed Model Repeated Measures Analysis — Unadjusted p-value; Mean difference(Mepolizumab 300-Placebo) = -0.4, 95% CI 2-sided [-1.5 to 0.8] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) collected from the start of study participation until the end of follow up (up to Week 60). On-treatment non-serious adverse events (AEs) reported from start of study treatment until 4 weeks after last dose.
Description: AEs and SAEs were collected in Safety Population which comprised of all randomized participants who received at least one dose of study treatment
Arm/Group | Placebo | Mepolizumab 100 mg SC | Mepolizumab 300 mg SC
All-Cause Mortality (participants affected / at risk) | 9/226 | 4/223 | 8/225
Serious Adverse Events (participants affected / at risk) | 68/226 | 57/223 | 60/225
Other Adverse Events (participants affected / at risk) | 137/226 | 147/223 | 137/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=226) | Mepolizumab 100 mg SC (N=223) | Mepolizumab 300 mg SC (N=225)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 37 (52) | 25 (34) | 32 (54)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 18 (19) | 16 (21) | 15 (16)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 5 (6) | 1 (1) | 3 (4)
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (6) | 3 (3) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=226) | Mepolizumab 100 mg SC (N=223) | Mepolizumab 300 mg SC (N=225)
Nasopharyngitis (Infections and infestations) | 48 (65) | 39 (57) | 40 (52)
Upper respiratory tract infection (Infections and infestations) | 20 (27) | 16 (19) | 12 (15)
Pneumonia (Infections and infestations) | 8 (9) | 10 (13) | 10 (11)
Bronchitis (Infections and infestations) | 8 (8) | 8 (12) | 11 (15)
Sinusitis (Infections and infestations) | 7 (11) | 8 (11) | 7 (9)
Influenza (Infections and infestations) | 11 (11) | 6 (7) | 3 (3)
Oral candidiasis (Infections and infestations) | 5 (7) | 3 (3) | 8 (9)
Rhinitis (Infections and infestations) | 5 (6) | 7 (9) | 4 (4)
Urinary tract infection (Infections and infestations) | 7 (8) | 7 (8) | 1 (1)
Injection site reaction (General disorders) | 10 (17) | 6 (6) | 11 (27)
Pyrexia (General disorders) | 9 (9) | 6 (7) | 12 (17)
Non-cardiac chest pain (General disorders) | 7 (7) | 5 (8) | 7 (8)
Fatigue (General disorders) | 4 (4) | 6 (6) | 8 (8)
Oedema peripheral (General disorders) | 3 (3) | 7 (7) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 14 (14) | 16 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 12 (14) | 10 (17)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 15 (15) | 11 (13)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 8 (12) | 10 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 15 (18) | 17 (21)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 10 (10) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (7) | 6 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 13 (16) | 8 (12)
Constipation (Gastrointestinal disorders) | 10 (10) | 7 (8) | 5 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (10) | 9 (13)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 9 (9) | 5 (5)
Headache (Nervous system disorders) | 20 (29) | 34 (62) | 22 (39)
Hypertension (Vascular disorders) | 3 (3) | 8 (9) | 7 (7)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.